CLINICAL TRIAL: NCT01415570
Title: Malnutrition, Diet and Racial Disparities in Chronic Kidney Disease (CKD) - A Prospective Data Collection Study
Brief Title: Malnutrition, Diet and Racial Disparities in Chronic Kidney Disease (CKD)
Acronym: MADRAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Davita Clinical Research (Industry)
Responsible Party: Sponsor
Other Study IDs: 14100; K24DK091419 (NIH)
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Kidney Disease (CKD); End-Stage Renal Disease (ESRD)
Keywords: Protein-energy wasting (PEW); racial disparities; hemodialysis; survival paradoxes; Stage 5
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic Hemodialysis Patients: Adult hemodialysis patients
- Chronic hemodialysis patients: Adult hemodialysis patients

SUMMARY:
In the United States, African Americans are 3.6 time and Hispanics 1.5 times more likely to suffer from chronic kidney disease and need dialysis treatment for life, when compared to the non-Hispanic Whites. Unfortunately many dialysis patients die, so that after 5 years only less than 35% are still alive. Dialysis patients who appear malnourished or who have muscle and fat wasting are even more likely to die. Interestingly, among dialysis patients, minorities (African Americans, Hispanics and Asian Americans) usually survive longer than the non-Hispanic Whites. If the investigators can discover the reasons for these so-called "racial survival disparities" of dialysis patients, the investigators may be able to improve survival for all dialysis patients and maybe even for many other people who suffer from other chronic diseases. During this 5 year study the investigators would like to test if a different nutrition and diet can explain better survival of minority dialysis patients. The investigators will also test if in additional to nutrition there are 2 other reasons for better survival of minority dialysis patients, namely differences in bone and minerals and differences in social and psychological and mental health. The investigators plan to study 450 hemodialysis patients every 6 months in several dialysis clinics in Los Angeles South Bay area. These subjects will include 30% African Americans, 30% Hispanics, 30% non-Hispanic Whites and 10% Asians. Every 6 months the investigators will examine their nutritional conditions, dietary intake, psycho-social conditions and quality of life, and will recruit 75 new subjects to replace those who left our study as a result of kidney transplantation, death or other reasons. Hence, the investigators estimate studying a total of 1,050 hemodialysis patients over 5 years. Clinical events such as hospital admissions and survival will be followed. Blood samples will be obtained every 6 months for measurements of hormones and "biomarkers", and the remainder of the blood will be stored in freezers for future measurements. The investigators plan to design and develop race and ethnicity specific nutritional risk scores and food questionnaires and will test some of these scores in larger national databases of hemodialysis patients. Almost a year after the study starts, the investigators also plan to do additional tests of body composition and dietary intake in a smaller group of these patients at the GCRC.

DETAILED DESCRIPTION:
I. SPECIFIC AIMS & HYPOTHESES I.1.HYPOTHESES: Despite higher burden of chronic kidney disease (CKD) in minorities, they have greater survival compared to non-Hispanic Whites with CKD. The investigators hypothesize that survival advantages of minority CKD patients (pts) result from biologically plausible mechanisms related to differences in nutritional status & diet (main hypothesis) or differences in bone-&-minerals and/or psychosocial & coping status (2 alternative hypotheses). Differences in these conditions may lead to different degrees of protein-energy wasting, inflammation, oxidative stress, & platelet activation, leading to thrombo-embolic & cardiovascular (CV) events. Discovering the biology of CKD racial survival disparities may lead to improving outcomes in both CKD and others chronic diseases.

During this 5-year study the principal investigator (Dr. Kalantar-Zadeh) will also help a number of early-career investigators to design and develop additional studies including research in minority populations with chronic diseases using data and resources of this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-85 yrs) patients
* HD > 4 weeks

Exclusion Criteria:

* Terminal disease with life expectancy < 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (18-85 yrs) patients, hemodialysis (HD) > 4 weeks
Sampling Method: Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2011-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 5-years (60 months)

SECONDARY OUTCOMES:
Quality of life | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kamyar Kalantar-Zadeh, MD, MPH, PhD, Principal Investigator — LABioMed at Harbor-UCLA
Locations (1):
- Harold Simmons Center for Kidney Disease Research & Epidemiology, Torrance, California, United States

REFERENCES:
- [Background] Noori N, Kovesdy CP, Dukkipati R, Feroze U, Molnar MZ, Bross R, Nissenson AR, Kopple JD, Norris KC, Kalantar-Zadeh K. Racial and ethnic differences in mortality of hemodialysis patients: role of dietary and nutritional status and inflammation. Am J Nephrol. 2011;33(2):157-67. doi: 10.1159/000323972. Epub 2011 Feb 4. PMID 21293117
- [Background] Feroze U, Noori N, Kovesdy CP, Molnar MZ, Martin DJ, Reina-Patton A, Benner D, Bross R, Norris KC, Kopple JD, Kalantar-Zadeh K. Quality-of-life and mortality in hemodialysis patients: roles of race and nutritional status. Clin J Am Soc Nephrol. 2011 May;6(5):1100-11. doi: 10.2215/CJN.07690910. Epub 2011 Apr 28. PMID 21527646
- [Background] Kalantar-Zadeh K, Kovesdy CP, Bross R, Benner D, Noori N, Murali SB, Block T, Norris J, Kopple JD, Block G. Design and development of a dialysis food frequency questionnaire. J Ren Nutr. 2011 May;21(3):257-62. doi: 10.1053/j.jrn.2010.05.013. Epub 2010 Sep 15. PMID 20833073
- [Background] Bross R, Noori N, Kovesdy CP, Murali SB, Benner D, Block G, Kopple JD, Kalantar-Zadeh K. Dietary assessment of individuals with chronic kidney disease. Semin Dial. 2010 Jul-Aug;23(4):359-64. doi: 10.1111/j.1525-139X.2010.00743.x. Epub 2010 Jul 29. PMID 20673254
- [Background] Bross R, Chandramohan G, Kovesdy CP, Oreopoulos A, Noori N, Golden S, Benner D, Kopple JD, Kalantar-Zadeh K. Comparing body composition assessment tests in long-term hemodialysis patients. Am J Kidney Dis. 2010 May;55(5):885-96. doi: 10.1053/j.ajkd.2009.12.031. Epub 2010 Mar 25. PMID 20346558
- [Background] Kalantar-Zadeh K, Kovesdy CP, Derose SF, Horwich TB, Fonarow GC. Racial and survival paradoxes in chronic kidney disease. Nat Clin Pract Nephrol. 2007 Sep;3(9):493-506. doi: 10.1038/ncpneph0570. PMID 17717562
- [Background] Kalantar-Zadeh K, Golan E, Shohat T, Streja E, Norris KC, Kopple JD. Survival disparities within American and Israeli dialysis populations: learning from similarities and distinctions across race and ethnicity. Semin Dial. 2010 Nov-Dec;23(6):586-94. doi: 10.1111/j.1525-139X.2010.00795.x. PMID 21175833
- [Background] Streja E, Kovesdy CP, Molnar MZ, Norris KC, Greenland S, Nissenson AR, Kopple JD, Kalantar-Zadeh K. Role of nutritional status and inflammation in higher survival of African American and Hispanic hemodialysis patients. Am J Kidney Dis. 2011 Jun;57(6):883-93. doi: 10.1053/j.ajkd.2010.10.050. Epub 2011 Jan 15. PMID 21239093
- [Background] Molnar MZ, Streja E, Kovesdy CP, Budoff MJ, Nissenson AR, Krishnan M, Anker SD, Norris KC, Fonarow GC, Kalantar-Zadeh K. High platelet count as a link between renal cachexia and cardiovascular mortality in end-stage renal disease patients. Am J Clin Nutr. 2011 Sep;94(3):945-54. doi: 10.3945/ajcn.111.014639. Epub 2011 Aug 3. PMID 21813809
- [Derived] Rhee CM, You AS, Nguyen DV, Brunelli SM, Budoff MJ, Streja E, Nakata T, Kovesdy CP, Brent GA, Kalantar-Zadeh K. Thyroid Status and Mortality in a Prospective Hemodialysis Cohort. J Clin Endocrinol Metab. 2017 May 1;102(5):1568-1577. doi: 10.1210/jc.2016-3616. PMID 28324018